CLINICAL TRIAL: NCT01395069
Title: Randomized Clinical Trial Comparing Prophylactic Nepafenac 0.1% and Ketorolac 0.5% Versus Placebo in Preventing Postoperative Macular Edema After Uncomplicated Phacoemulsification Cataract Extraction (PNK)
Brief Title: Prophylactic Nepafenac and Ketorolac Versus Placebo in Patients Undergoing Cataract Surgery
Acronym: PNK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Sherif R El-Defrawy, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PNK
Record Dates: First submitted 2011-07-11; First posted 2011-07-15 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Macular Edema
Keywords: Post-cataract surgery; macular edema
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nepafenac 0.1% (Active Comparator)
  Interventions: Drug: Nepafenac 0.1%
- Ketorolac 0.5% (Active Comparator)
  Interventions: Drug: Ketorolac 0.5%
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo (sterile saline drops)

INTERVENTIONS:
Drug: Nepafenac 0.1% — 1 drop QID for 1 month
  Arms: Nepafenac 0.1%
Drug: Ketorolac 0.5% — 1 drop QID for 1 month
  Arms: Ketorolac 0.5%
Other: Placebo (sterile saline drops) — 1 drop QID for 1 month
  Arms: Placebo

SUMMARY:
Assess prophylactic efficacy of topical non-steroidal anti-inflammatory drops in preventing macular edema. Patient undergoing uncomplicated cataract surgery will be enrolled and randomized to nepafenac, ketorolac, or placebo. Follow-up will occur at 1 month with ocular coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Age 18 years and older

Exclusion Criteria:

* Any pre-existing retinal disease (e.g., diabetic retinopathy, vein occlusion, exudative macular degeneration, etc.)
* Previous uveitis
* Previous intraocular surgery
* Allergy or hypersensitivity to NSAIDs
* Complicated cataract surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2010-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change in macular volume (as quantified by OCT) at one month (compared to baseline) | baseline and one month after surgery

SECONDARY OUTCOMES:
COMTOL health-related quality-of-life | one month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sherif El-Defrawy, MD PhD, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada